CLINICAL TRIAL: NCT05572229
Title: A Phase 2 Study of Teclistamab in Combination With Daratumumab or Lenalidomide in Elderly Patients With Newly Diagnosed Multiple Myeloma
Brief Title: Study of Teclistamab in Combination in Elderly Patients With Multiple Myeloma
Acronym: IFM2021-01
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2022_0174; 2022-001594-31 (EudraCT Number)
Record Dates: First submitted 2022-09-27; First posted 2022-10-07 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Multiple Myeloma
Keywords: Newly diagnosed Multiple Myeloma; Elderly patients; Teclistamab; Daratumumab; Lenalidomide; Toxicity
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tec-Dara (Experimental): For patients assigned to cohort A (Tec-Dara) patients will receive Tec-Dara until documented PD or unacceptable toxicity
  Interventions: Drug: Teclistamab; Drug: Daratumumab
- Tec-Len (Experimental): For patients assigned to cohort B (Tec-Len) patients will receive Tec-Len until documented PD or unacceptable toxicity
  Interventions: Drug: Teclistamab; Drug: Lenalidomide

INTERVENTIONS:
Drug: Teclistamab — Teclistamab will be administered via a subcutaneous injection (SC)
  Other Names: JNJ-64007957
Drug: Daratumumab — Daratumumab will be administered via a subcutaneous injection (SC)
  Arms: Tec-Dara
Drug: Lenalidomide — Lenalidomide will be administered orally
  Arms: Tec-Len

SUMMARY:
The primary hypothesis of this study is that teclistamab SC in combination with daratumumab SC or lenalidomide will be safe and induce a high rate of VGPR or better in newly diagnosed multiple myeloma patients

This is an open-label, multicenter, non-comparative, 2-cohort, 2-stage with interruption of enrollment for an efficacy and safety interim analysis, interventional Phase 2 study evaluating the efficacy and safety of a combination with Tec-Dara (Cohort A) or Tec-Len (Cohort B) in patients with newly diagnosed multiple myeloma who are not eligible for SCT.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be at least ≥65 years of age at the time of informed consent with documented multiple myeloma as defined by the criteria below:

   Multiple myeloma diagnosis according to IMWG diagnostic criteria

   Measurable disease at Screening as defined by any of the following:

   Serum monoclonal paraprotein (M-protein) level ³ 0.5 g/dL; or Urine M protein level ³ 200 mg/24 hours; or Serum Ig FLC ³ 10 mg/dL and abnormal serum Ig kappa/lambda FLC ratio
2. Have an ECOG performance status score of 0-2
3. Not considered for high-dose chemotherapy and autologous SCT
4. Have clinical laboratory values meeting the criteria during the Screening Phase.
5. A male patient must wear a condom (with spermicidal foam/gel/film/cream/suppository) when engaging in any activity that allows for passage of ejaculate to another person during the study and for a minimum of 4 weeks after the last dose of lenalidomide or for a period of 3 months after the last dose of other study treatments, whichever occurs later. If the male patient's partner is a female of childbearing potential, she must also be practicing a highly effective method of contraception. If the male patient is vasectomized, he still must wear a condom (with or without spermicidal foam/gel/film/cream/suppository), but his female partner is not required to use contraception.

7. A male patient must agree not to donate sperm for the purpose of reproduction during the study and for a minimum of 4 weeks after the last dose of lenalidomide or for period of 3 months after receiving the last dose of other study treatments, whichever occurs later.

8. Must sign an ICF (or their legally acceptable representative must sign in accordance with local requirements) indicating that the patient understands the purpose of, and procedures required for, the study and is willing to participate in the study.

9. Must be willing and able to adhere to the lifestyle restrictions specified in this protocol.

Exclusion Criteria:

Medical Conditions

1. CNS involvement or clinical signs of meningeal involvement of multiple myeloma. If either is suspected, negative whole brain MRI and lumbar cytology are required.
2. Plasma cell leukemia, Waldenström's macroglobulinemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, M-protein, and skin changes), or primary light chain amyloidosis.
3. Any ongoing myelodysplastic syndrome or B cell malignancy (other than multiple myeloma).
4. Any history of malignancy, other than multiple myeloma, which is considered at high risk of recurrence requiring systemic therapy
5. Any active malignancies (ie, progressing or requiring treatment change in the last 24 months) other than multiple myeloma.
6. Stroke, transient ischemic attack, or seizure within 6 months prior to signing ICF.
7. Presence of the a cardiac conditions.

   Tec-Dara-specific
8. COPD with a FEV1 <50% of predicted normal. Note that FEV1 testing is required for patients with known or suspected of having COPD or asthma and patients must be excluded if FEV1 <50% of predicted normal.
9. Moderate or severe persistent asthma within the past 2 years or uncontrolled asthma of any classification. Note that FEV1 testing is required for patients known or suspected asthma and patients must be excluded if FEV1 <50% of predicted normal.

   Prior/Concomitant Therapy
10. Radiotherapy within 14 days or focal radiation within 7 days.
11. Received a cumulative dose of corticosteroids equivalent to ≥140 mg of prednisone within 14-days before the first dose of study drug (does not include pretreatment medications).
12. Received a live, attenuated vaccine within 4 weeks before the first dose of study drug. Non-live or non-replicating vaccines authorized for emergency use (eg, COVID-19) are allowed.
13. Any prior therapy for multiple myeloma or smoldering myeloma other than a short course of corticosteroids prior to signing ICF (not to exceed 40 mg of dexamethasone, or equivalent per day for a maximum of 4 days, total of 160 mg dexamethasone or equivalent).
14. Contraindications or life-threatening allergies, hypersensitivity, or intolerance to any study drug or its excipients.

    Diagnostic Assessments
15. HIV positive.
16. Hepatitis B infection.
17. Active hepatitis C infection as measured by positive HCV-RNA testing. Other Exclusions
18. Women of childbearing potential
19. Patient had major surgery or had significant traumatic injury within 2 weeks prior to the start of administration of study treatment, or will not have fully recovered from surgery., or has major surgery planned during the time the patient is expected to be treated in the study or within 2 weeks after administration of the last dose of study treatment.
20. Concurrent medical or psychiatric condition or disease that is likely to interfere with study procedures or results.
21. Patient plans to father a child while enrolled in this study or within 3 months after the last dose of study intervention.
22. Person under guardianship, trusteeship or deprived of freedom by a judicial or administrative decision.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2023-12-21 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Rate of very good partial response (VGPR) or better according to the IMWG criteria in patients with newly diagnosed multiple myeloma after 4 cycles of treatment with Tec-Dara or Tec-Len | At the end of 4 th cycle (each cycle is 28 days), an average 4 months

SECONDARY OUTCOMES:
Treatment-emergent adverse events according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE, Version 5.0). | From date of randomization until the date of first documented progression,assessed up to 5 years
Overall response rate(PR or better) as defined by the IMWG response criteria | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years
Very good partial response or better, defined as VGPR or CR according to the IMWG criteria at the time of data cutoff | TFrom date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years
Complete response or better, defined as negative immunofixation of serum and urine, and disappearance of any soft tissue plasmacytomas, and <5% plasma cells in bone marrow* | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years
Time to response | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years
Duration of response | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years
Time from randomization to discontinuation of therapy for any reason including death, progression or toxicity | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years
Overall survival time | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years
  OS, measured from the date of the first dose of study treatment to the date of the patient's death. If the patient is alive or the vital status is unknown at last contact, then the patient's data will be censored at the date the patient was last known to be alive
TTTF, defined as the time from the date of the first dose of study treatment to discontinuation of therapy for any reason including death, progression, toxicity | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years
TTNT, defined as the time from date of the first dose of study treatment to the start of the next-line treatmentTime-to-next treatment | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years
Rate of minimal residual disease (MRD)-negativity (at level of 10-5 and 10-6 by NGS) at 6 months | at 6 months
Rate of Sustained MRD-negativity-(at level of 10-5 and 10-6 by NGS) | at 18 months (12 months after the initial MRD time point).

CONTACTS AND LOCATIONS:
Overall Officials: Salomon MANIER, MD, Principal Investigator — University Hospital, Lille
Locations (29):
- France (29):
  - Chu Amiens - Hopital Sud, Amiens
  - Chru Angers, Angers
  - Ch D'Avignon, Avignon
  - Centre Hospitalier de La Cote Basque, Bayonne
  - Chu de Besancon, Besançon
  - Aphp Hopital Avicenne, Bobigny
  - Chu de Caen, Caen
  - Chu Dijon Bourgogne, Dijon
  - Ch de Dunkerque, Dunkirk
  - Chu de Grenoble, La Tronche
  - Centre Hospitalier de Versailles, Le Chesnay
  - Chu de Lille, Hopital Claude Huriez, Lille
  - Chu Limoges, Limoges
  - Centre Leon Berard, Lyon
  - Chr Metz-Thionville, Metz
  - Chu Montpellier, Montpellier
  - Hopital E. Muller- Ghrmsa, Mulhouse
  - Chru de Nancy, Hopitaux de Brabois, Nancy
  - Chu de Nantes Site Hotel Dieu, Nantes
  - Aphp - Chu Henri Mondor, Paris
  - Aphp - Hopital Saint Antoine, Paris
  - Aphp - Hopital Saint Louis, Paris
  - Chu Bordeaux, Pessac
  - Chu de Poitiers, Poitiers
  - Chu de Reims, Reims
  - Chu Pontchaillou, Rennes
  - Hopitaux Universitaire de Strasbourg - Hopital Hautepierre, Strasbourg
  - Oncopole Chu Toulouse, Toulouse
  - Chru Bretonneau, Tours